CLINICAL TRIAL: NCT00739830
Title: A Randomized Phase II Trial of Ridaforolimus (AP23573; MK-8669) Compared to Progestin or Chemotherapy in Female Adult Patients With Advanced Endometrial Carcinoma
Brief Title: Clinical Trial of Ridaforolimus Compared to Progestin or Chemotherapy for Advanced Endometrial Carcinoma (MK-8669-007 AM6)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-007; AP23573-07-205 (Other: ARIAD study number)
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — ridaforolimus; Medroxyprogesterone Acetate; Megestrol Acetate; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 40 mg once daily oral tablets for 5 days followed by 2 days without ridaforolimus
  Interventions: Drug: ridaforolimus
- 2 (Active Comparator): Investigator's choice of: oral medroxyprogesterone acetate tablets 200 mg daily or oral megestrol acetate tablets 40 mg 4 times per day (160 mg daily) OR Chemotherapy - carboplatin, paclitaxel, doxorubicin, pegylated liposomal doxorubicin or topotecan administered as a single agent or as a doublet, and will be administered at doses and schedules chosen by the investigator
  Interventions: Drug: medroxyprogesterone acetate tablets OR megestrol acetate; Drug: chemotherapy

INTERVENTIONS:
Drug: ridaforolimus — 40 mg once daily oral tablets for 5 days followed by 2 days without ridaforolimus
  Other Names: deforolimus, AP23573, MK-8669; ridaforolimus was also known as deforolimus until May 2009
  Arms: 1
Drug: medroxyprogesterone acetate tablets OR megestrol acetate — oral medroxyprogesterone acetate tablets 200 mg daily OR oral megestrol acetate tablets 40 mg 4 times per day (160 mg daily)
  Arms: 2
Drug: chemotherapy — Chemotherapy - carboplatin, paclitaxel, doxorubicin, pegylated liposomal doxorubicin or topotecan administered as a single agent or as a doublet, and will be administered at doses and schedules chosen by the investigator
  Arms: 2

SUMMARY:
The purpose of this study is to compare progression-free survival (PFS) of patients with advanced, recurrent or metastatic endometrial cancer who have received one, but not more than two, prior lines of chemotherapy either as adjuvant therapy or treatment for advanced disease, and then when treated with ridaforolimus or the investigators' choice of progestin or chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Endometrial cancer
* Patients must have been treated with at least one line of chemotherapy, but not more than two lines of chemotherapy, and experienced progressive disease
* At least one measurable lesion
* ECOG performance status less than or equal to 1
* Minimum life expectancy of 3 months
* Adequate renal and hepatic function
* Adequate bone marrow function
* Serum cholesterol <350 mg/dL and triglycerides < 400 mg/dL
* Able to understand and give written informed consent
* Females of childbearing potential must have a negative pregnancy test and use approved contraception from screening to 30 days after the last study drug is given

Exclusion Criteria:

* Two lines of chemotherapy for recurrent or metastatic disease
* Chemotherapy for recurrent or metastatic disease administered within six months of adjuvant therapy
* More than two lines of chemotherapy of any type
* Prior therapy with hormonal agents
* Women who are pregnant or lactating
* Presence of brain or other central nervous system metastases
* Prior therapy with rapamycin, rapamycin analogues or tacrolimus or known sensitivity to these agents
* Anticancer treatment (chemotherapy, radiotherapy) within 4 weeks prior to randomization
* Ongoing toxicity associated with prior anticancer therapy
* Inadequate recovery from any prior surgical procedure or having undergone any major surgical procedure within 2 weeks prior to randomization.
* Another primary malignancy within the past five years (except for non-melanoma skin cancer and cervical carcinoma in situ)
* Known Grade 3 or 4 hypersensitivity to macrolide antibiotics
* Significant uncontrolled cardiovascular disease
* Active infection
* Known HIV infection
* Known Hepatitis B or C infection
* Newly diagnosed (within 3 months before enrollment) or poorly controlled Type 1 or 2 diabetes
* Concurrent treatment with immunosuppressive agents
* A requirement for concurrent treatment with medication that strongly induce or inhibit cytochrome P450 (CYP3A)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-08; Primary Completion 2011-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization up to 30 months

SECONDARY OUTCOMES:
The proportion of patients progression free at 16 weeks as assessed using modified RECIST guidelines. | From randomization to Week 16
The proportion of patients progression free at 26 weeks as assessed using modified RECIST guidelines | From randomization to Week 26
Overall survival | From randomization up to 30 months
Best target lesion response, defined as best change in sum of the target lesions from baseline to disease progression | From randomization up to 30 months
Safety and tolerability | From randomization up to 30 days after discontinuation of treatment

REFERENCES:
- [Background] Oza AM, Pignata S, Poveda A, McCormack M, Clamp A, Schwartz B, Cheng J, Li X, Campbell K, Dodion P, Haluska FG. Randomized Phase II Trial of Ridaforolimus in Advanced Endometrial Carcinoma. J Clin Oncol. 2015 Nov 1;33(31):3576-82. doi: 10.1200/JCO.2014.58.8871. Epub 2015 Jun 15. PMID 26077241